CLINICAL TRIAL: NCT05726760
Title: Observational Study of Peripheral Skin Temperature Changes Following Spinal Anaesthesia for Category 4 Lower Segment Caesarean Section (LSCS)
Brief Title: Peripheral Skin Temperature Changes Following Spinal Anaesthesia for Category 4 LSCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Obstetric Anaesthetists' Association United Kingdom (Other)
Responsible Party: Principal Investigator, Dr Laura Kessack, Consultant Anaesthetist, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: IRAS263967
Record Dates: First submitted 2021-08-21; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group - Parturients having spinal anaesthesia: ASA 1 and 2 full term (37-42 weeks), parturients with singleton pregnancy, normal placental position, scheduled for category 4 LSCS under 'single-shot' spinal anaesthesia will be recruited. The investigators intend to recruit 60 parturients. The parturients will undergo an informed consent process including an explanation of the methods and risks of the study. A patient information leaflet will be provided for the parturients.
  Interventions: Behavioral: Seeking informed consent for participation in the study.; Device: Temperature measurement by Braun Welch Allyn tympanic membrane thermometer device to the dorsum of the right and left feet above space between the 2nd and 3rd metatarsal bones.; Device: Covidien Mon-a-Therm skin temperature probes will be applied to the dorsum of the right and left feet above space between the 2nd and 3rd metatarsal bones.; Device: Temperature measurement by Braun Welch Allyn tympanic membrane thermometer device to the ear.
- Control group - Parturients not having spinal anaesthesia: 6 parturients will be recruited as a control group. ASA 1 and 2 full term (37-42 weeks), parturients with singleton pregnancy, normal placental position, scheduled for category 4 LSCS under 'single-shot' spinal anaesthesia will be recruited.
  Interventions: Behavioral: Seeking informed consent for participation in the study.; Device: Temperature measurement by Braun Welch Allyn tympanic membrane thermometer device to the dorsum of the right and left feet above space between the 2nd and 3rd metatarsal bones.; Device: Covidien Mon-a-Therm skin temperature probes will be applied to the dorsum of the right and left feet above space between the 2nd and 3rd metatarsal bones.; Device: Temperature measurement by Braun Welch Allyn tympanic membrane thermometer device to the ear.

INTERVENTIONS:
Behavioral: Seeking informed consent for participation in the study. — The parturients will undergo an informed consent process including an explanation of the methods and risks of the study. The Anaesthetist or researcher will conduct this process. A patient information leaflet will be provided for the parturients.
Device: Temperature measurement by Braun Welch Allyn tympanic membrane thermometer device to the dorsum of the right and left feet above space between the 2nd and 3rd metatarsal bones. — The Anaesthetist or researcher and recovery nurse will conduct the intervention in theatre and in the recovery ward.
Device: Covidien Mon-a-Therm skin temperature probes will be applied to the dorsum of the right and left feet above space between the 2nd and 3rd metatarsal bones. — The Anaesthetist or researcher will conduct the intervention in theatre. The probes will be removed in the recovery ward.
Device: Temperature measurement by Braun Welch Allyn tympanic membrane thermometer device to the ear. — The Anaesthetist or researcher and recovery nurse will conduct the intervention in theatre and in the recovery ward.

SUMMARY:
Regional anaesthesia of the lower limbs blocks sympathetic nerve fibres as well as sensory and motor fibres. It has been documented previously in the non-pregnant population that the blockade of sympathetic nerve fibres by regional anaesthesia (including spinal, epidural and lumbar plexus anaesthesia) results in vasodilation of peripheral blood vessels and an increase in the blood flow to the skin, increasing the peripheral skin temperature. Additionally thermoregulation has been found to be impaired more by spinal anaesthesia than epidural anaesthesia. The aim of the study is to measure peripheral skin temperature changes occurring in the lower limbs following spinal anaesthesia in the pregnant obstetric population undergoing category 4 lower segment caesarean section. The hypothesis is that peripheral skin temperature will rise following spinal anaesthesia and that this temperature change could be used as a measure of bilateral sympathetic block which may be an indicator of potential success of spinal anaesthesia. Future follow up studies could then potentially determine if peripheral skin temperature can also be used as a marker to determine the success of epidural analgesia for labour.

The study will involve temperature measurement by Covidien Mon-a-Therm skin temperature probes and Braun Welch Allyn tympanic membrane thermometer devices on the dorsum of the right and left feet. The study will last from the time the parturient arrives in theatre for their lower segment caesarean section until the parturient leaves the recovery area.

DETAILED DESCRIPTION:
The hypothesis is that peripheral skin temperature will rise following spinal anaesthesia and that this temperature change could be used as an indicator of potential success of spinal anaesthesia.

This is an observational study. The investigators will obtain ethics committee approval for conducting the study. ASA 1 and 2 full term (37-42 weeks), parturients with singleton pregnancy, normal placental position, scheduled for category 4 LSCS under 'single-shot' spinal anaesthesia will be recruited. The investigators intend to recruit 60 parturients. The parturients will undergo an informed consent process including an explanation of the methods and risks of the study. A patient information leaflet will be provided for the parturients.

The data will be collected on a password protected spread-sheet with no patient identifiable information. A grant for funding has been granted from the Obstetric Anaesthetists' Association.

Prior to establishment of spinal anaesthesia, the skin temperature of the parturient's feet will be measured on the dorsum of the right and left feet above space between the 2nd and 3rd metatarsal bones while the parturient is lying supine with left lateral tilt. The temperature will be measured by Covidien Mon-a-Therm skin temperature probes and a Braun Welch Allyn tympanic membrane thermometer device. Following spinal injection when the parturient is lying supine with lateral tilt, the temperature will be re-measured by Covidien Mon-a-Therm skin temperature probes and a Braun Welch Allyn tympanic membrane thermometer device. The skin temperature of the parturient's feet will be monitored continuously by the Covidien Mon-a-Therm skin temperature probes using the GE Healthcare monitor with readings transcribed every 1 minute by the research investigator until transfer onto the bed at the end of surgery. The skin temperature of the parturient's feet will be measured and recorded every 1 minute using a Braun Welch Allyn tympanic membrane thermometer device until the sterile drapes are applied prior to commencing the operation and then again after removal of the drapes prior to transfer onto the bed. Following transfer to the post-operative recovery area, the skin temperature of the parturient's feet will be measured and recorded every 10 minutes using a Braun Welch Allyn tympanic membrane thermometer device until discharged to the ward from the recovery area (usually 2 hours from departmental guidelines).

Theatre room temperature will be measured and recorded at the start of anaesthesia and at the end of surgery using a room thermometer. Surgical drapes will be applied over the parturient's lower limbs during the caesarean section procedure as per the investigators routine practice. The ambient temperature under the surgical drapes will be measured and recorded at the start of anaesthesia and at the end of surgery using a room thermometer.

Tympanic temperature will be measured by a Braun Welch Allyn tympanic membrane thermometer device before spinal anaesthesia and then every 30 minutes until the end of surgery as per NICE clinical guideline 65.

Spinal anaesthesia will be conducted as per usual practice. All intravenous fluids will be given through a fluid warmer.

Parturient data to be recorded will include: Age, Weight, Height, BMI, total dose of intra-operative vasopressor given, highest estimated dermatome level of anaesthesia to cold (ethyl chloride spray) bilaterally prior to commencing surgery, level motor block using straight leg raise as per normal practice when anaesthesia ready for surgery, duration of surgery, estimated blood loss, total volume of intravenous fluids given (including any blood products). Dermatome level of anaesthesia will be measured to cold (ethyl chloride spray) level and motor block will be measured using straight leg raise as per normal practice, in recovery, every 30 minutes.

6 parturients will be recruited as a control group. The skin temperature of these parturient's feet will be measured on the dorsum of the right and left feet above space between the 2nd and 3rd metatarsal bones while the parturient is lying supine with left lateral tilt in theatre. The temperature will be measured by Covidien Mon-a-Therm skin temperature probes and a Braun Welch Allyn tympanic membrane thermometer device. The sterile drapes will be applied and the skin temperature of the parturient's feet will be monitored continuously by the Covidien Mon-a-Therm skin temperature probes using the GE Healthcare monitor with readings transcribed every 1 minute by the research investigator for 30 minutes. After 30 minutes, the skin temperature of the parturient's feet will be measured and recorded every 1 minute using a Braun Welch Allyn tympanic membrane thermometer device for 5 minutes. Theatre room temperature will be measured and recorded for this control group of parturients. The ambient temperature under the surgical drapes will be measured and recorded using a room thermometer.

Inclusions / exclusions:

Parturients will be excluded from the study if the parturient refuses or if they have medical conditions that may affect peripheral temperature and therefore the results of the study. The exclusion criteria are: Parturients converted to other forms of anaesthesia (not just spinal anaesthesia); Parturients with a pyrexia / sepsis; Parturients with peripheral vascular disease (including Raynauds); Parturients with cardiovascular disease; Parturients with diabetes mellitus (gestational, type 1 or 2); Hypertensive disorders of pregnancy; ASA 3+ Parturients; BMI >40 or <18; Parturient refusal.

ELIGIBILITY:
Inclusion Criteria:

* Full term (37-42 weeks) parturients
* ASA 1 and 2
* Singleton pregnancy
* Normal placental position
* Scheduled for category 4 LSCS
* 'Single-shot' spinal anaesthesia
* Signed informed consent
* Received a patient information leaflet

Exclusion Criteria:

* Any medical conditions that may affect peripheral temperature
* Parturients converted to other forms of anaesthesia (not just spinal anaesthesia)
* Parturients with a pyrexia / sepsis
* Parturients with peripheral vascular disease (including Raynauds)
* Parturients with cardiovascular disease
* Parturients with diabetes mellitus (gestational, type 1 or 2)
* Parturients with hypertensive disorders of pregnancy
* ASA 3+ Parturients
* BMI >40 or <18
* Parturient refusal.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Study Population: ASA 1 and 2 full term (37-42 weeks), parturients with singleton pregnancy, normal placental position, scheduled for category 4 LSCS under 'single-shot' spinal anaesthesia will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2023-03-21 (Estimated); Study Completion 2023-05-21 (Estimated)

PRIMARY OUTCOMES:
The peripheral skin temperature of the dorsum of the feet measured prior to and following establishment of a spinal anaesthetic block in parturients undergoing category 4 caesarean section. | During the spinal anaesthetic inserted for the lower segment caesarean section in theatre
  Temperature measured on the dorsum of both feet.

SECONDARY OUTCOMES:
Measurement of peripheral temperature using the Infra red tympanic thermometer. | During the spinal anaesthetic and lower segment caesarean section in theatre and for the 2 hours the parturient is in the recovery area.
  Infra red tympanic thermometers measure the frequency of infrared light emitted by the tympanic membrane. The investigators propose that infra red tympanic thermometers could also be used to measure the frequency of infrared light emitted by the skin.
The peripheral skin temperature of the dorsum of the feet measured in recovery following establishment of a spinal anaesthetic block in parturients undergoing category 4 caesarean section. | During the 2 hours the parturient is in the recovery area.
  Temperature measured on the dorsum of both feet.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kessack, MBChB2003, Principal Investigator — Cambridge University Hospitals
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Werdehausen R, Braun S, Hermanns H, Freynhagen R, Lipfert P, Stevens MF. Uniform distribution of skin-temperature increase after different regional-anesthesia techniques of the lower extremity. Reg Anesth Pain Med. 2007 Jan-Feb;32(1):73-8. doi: 10.1016/j.rapm.2006.07.009. PMID 17196496
- [Background] Hermanns H, Werdehausen R, Hollmann MW, Stevens MF. Assessment of skin temperature during regional anaesthesia-What the anaesthesiologist should know. Acta Anaesthesiol Scand. 2018 Oct;62(9):1280-1289. doi: 10.1111/aas.13176. Epub 2018 Jun 25. PMID 29938773
- [Background] Park SY, Nahm FS, Kim YC, Lee SC, Sim SE, Lee SJ. The cut-off rate of skin temperature change to confirm successful lumbar sympathetic block. J Int Med Res. 2010 Jan-Feb;38(1):266-75. doi: 10.1177/147323001003800131. PMID 20233538
- [Background] Bengtsson M. Changes in skin blood flow and temperature during spinal analgesia evaluated by laser Doppler flowmetry and infrared thermography. Acta Anaesthesiol Scand. 1984 Dec;28(6):625-30. doi: 10.1111/j.1399-6576.1984.tb02134.x. PMID 6240882
- [Background] Penno A, Arumugam M, Antweiler G, Laubert T, Habermann J, Bruch HP. [Increase in skin surface temperature in spinal anesthesia. Predictive value for probability of surgical tolerance]. Anaesthesist. 2012 Sep;61(9):770-6. doi: 10.1007/s00101-012-2076-3. Epub 2012 Sep 8. German. PMID 22955888
- [Background] Jetzek-Zader M, Hermanns H, Freynhagen R, Lipfert P, Stevens MF. Increase in skin temperature after spinal anesthesia in infants. Reg Anesth Pain Med. 2006 Nov-Dec;31(6):519-22. doi: 10.1016/j.rapm.2006.07.007. PMID 17138194
- [Background] Ehrlich PF, Vedulla G, Cottrell N, Seidman PA. Monitoring intraoperative effectiveness of caudal analgesia through skin temperature variation. J Pediatr Surg. 2003 Mar;38(3):386-9. doi: 10.1053/jpsu.2003.50113. PMID 12632354
- [Background] Saito T, Sessler DI, Fujita K, Ooi Y, Jeffrey R. Thermoregulatory effects of spinal and epidural anesthesia during cesarean delivery. Reg Anesth Pain Med. 1998 Jul-Aug;23(4):418-23. doi: 10.1016/s1098-7339(98)90017-7. PMID 9690596
- [Background] Griffin RP, Reynolds F. The association between foot temperature and asymmetrical epidural blockade. Int J Obstet Anesth. 1994 Jul;3(3):132-6. doi: 10.1016/0959-289x(94)90224-0. PMID 15636935

DOCUMENTS (2):
  • Study Protocol (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT05726760/Prot_000.pdf
  • Informed Consent Form (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT05726760/ICF_001.pdf